CLINICAL TRIAL: NCT06953895
Title: The Immediate Effect of Mulligan's Mobilization With Movement on Shoulder Girdle' Pain, Range of Motion and Muscle Activity, in Subjects With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Daniela Ferreira Carneiro, MSc, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00853
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Subacromial impingement syndrome; Mobilization with movement; Pressure pain threshold; Surface electromyography
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Movement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The Mulligan's MWM group received mobilization with movement in the glenohumeral joint, as described by Mulligan. The participant was seated, and the physiotherapist was placed on the opposite side to the affected shoulder with the thenar eminence of one hand over the anterior aspect of the humeral head, and the other hand over the spine of the scapula posteriorly of the affected shoulder. The hand over the humeral head performed a posterolateral glide, while the other hand stabilized the scapula. This maneuver was sustained while the participant asked to raise the arm in scapular plan (as explained above) without pain. The physiotherapist previously determined the amount of posterolateral pressure which was the best to abolish the pain during shoulder scaption for each participant.
  Interventions: Procedure: Mulligan's Mobilization With Movement
- Placebo Group (Placebo Comparator): In the Placebo group, no effective intervention was performed, the participant was asked to raise the affected arm in scapular plane without pain, while the physiotherapist placed their hands-on shoulder, with the same manual contacts described in Mulligan's MWM group, but without performing any pressure.
  Interventions: Procedure: Active Mobilization

INTERVENTIONS:
Procedure: Mulligan's Mobilization With Movement — The Mulligan's MWM group received mobilization with movement in the glenohumeral joint, as described by Mulligan. The participant was seated, and the physiotherapist was placed on the opposite side to the affected shoulder with the thenar eminence of one hand over the anterior aspect of the humeral head, and the other hand over the spine of the scapula posteriorly of the affected shoulder. The hand over the humeral head performed a posterolateral glide, while the other hand stabilized the scapula. This maneuver was sustained while the participant asked to raise the arm in scapular plan (as explained above) without pain. The physiotherapist previously determined the amount of posterolateral pressure which was the best to abolish the pain during shoulder scaption for each participant. The participants performed three sets of 10 trials with a resting time of 30 seconds between each set. After intervention was allowed a resting time of three minutes.
  Other Names: MWM
  Arms: Intervention group
Procedure: Active Mobilization — In the Placebo group, no effective intervention was performed, the participant was asked to raise the affected arm in scapular plane without pain, while the physiotherapist placed their hands-on shoulder, with the same manual contacts described in Mulligan's MWM group, but without performing any pressure.
  The participants performed three sets of 10 trials with a resting time of 30 seconds between each set. After intervention was allowed a resting time of three minutes.
  Arms: Placebo Group

SUMMARY:
The aim of present study was to evaluate the immediate effect of Mulligan's mobilization with movement on shoulder girdle' pain, range of motion (ROM) and muscle activity, in subjects with shoulder impingement syndrome

DETAILED DESCRIPTION:
A randomized, single-blind, placebo-controlled clinical trial was conducted with a sample composed by twenty-four volunteers with SIS, divided in Mulligan's MWM and Placebo groups. Pain intensity in Neer impingement signal and Hawkins-Kennedy impingement test, pressure pain threshold (PPT) on the lateral aspect of shoulder, ROM of shoulder scaption until onset of pain, as well as the activity of trapezius (upper, middle and lower fibers) and serratus anterior muscles during this movement, were evaluated before and immediate (post-) intervention. The Mulligan's MWM group received a mobilization with movement technique in the glenohumeral joint (sustained posterolateral glide during shoulder scaption), while no effective intervention was performed in the Placebo group.

ELIGIBILITY:
Inclusion Criteria:

Participants had superolateral shoulder pain and two out of four specified objective signs and symptoms:

* positive Neer test;
* positive Hawkins-Kennedy test;
* painful limitation of active arm elevation (flexion, abduction, scaption);
* pain or limitation with functional movement patterns of hand behind back or hand behind head.

Exclusion Criteria:

* physician diagnosis of adhesive capsulitis;
* grade III rotator cuff tear;
* calcific tendinosis confirmed by radiology;
* systemic or neurological disorder;
* cervical radiculopathy; a history of shoulder surgery;
* corticosteroid injection within the past month;
* subjects who had received physical therapy intervention for their shoulder within the past three months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | baseline
  The participant was asked to rate the pain intensity in Neer impingement signal and Hawkins-Kennedy impingement test, using a 100 mm visual analogue scale.
Pain Pressure Threshold on the lateral aspect of shoulder | baseline
  Pressure algometry was performed to assess PPT on the lateral aspect of shoulder. A hand-held electronic pressure algometer Force One FDIX (Wagner Instruments, Greenwich CT, United States of America) with a 1 cm2 rubber-tipped probe area was applied perpendicular to the skin at a rate of 1 kg per second. The PPT was measured over the most sensitive point to manual palpation of the lateral aspect of shoulder. This region was marked with a permanent marker so that the same point could be used pre- and post-intervention. The researcher instructed the participant to say "ouch" as soon as sensation changed from feeling pressure to feeling pain. Three trials were performed, with a resting time of 30 seconds and a subsequent analysis of its average.
Shoulder ROM | baseline
  Photogrammetry was performed to assess ROM of shoulder scaption until onset of pain. The ROM was recorded by photography, using a digital camera (30 frames/ second) placed in a perpendicular position to the plane of motion, at a distance of 3 meters from a flat surface. The photography was subsequently analyzed by a postural analysis software (SAPo version 0.69, open source software). To ensure consistent reference points, spherical markers were placed on the skin: one over the acromion and the last over the lateral epicondyle. The participant was asked to raise the arm until feeling pain, with elbow fully extended and thumb pointed up along a flat vertical surface positioned 30º anterior to the frontal plane.
Shoulder muscle activity | baseline
  Surface electromyography (sEMG) was performed to assess the muscle activity of trapezius (upper, middle and lower) and SA, during concentric and eccentric phases of shoulder scaption. The muscle activity was recorded by BioPlux research device (Plux wireless biosignals S.A., Arruda dos Vinhos, Portugal) with 12-bit analog channels and a sampling frequency of 1000 Hz, using double differential electrode leads. To perform sEMG, the participant's hair was shaved, an abrasive cream was used to remove dead cells from the skin's surface, and the skin was cleaned with isopropyl alcohol (70%) to remove oil and remaining dead cells. An electrode impedance checker (Noraxon Corporate, Scottsdale AZ, United States of America) was used to ensure that impedance levels were less than 5 KΩ, which was considered to signify the satisfactory acquisition of the sEMG signal.

CONTACTS AND LOCATIONS:
Locations (1):
- E2S | P.PORTO - Escola Superior de Saúde do Politécnico do Porto, Porto, Porto District, Portugal